CLINICAL TRIAL: NCT04131439
Title: Role of Multislice Computed Tomography and Magnetic Resonance Imaging in Preoperative Cochlear Implant Evaluation
Brief Title: CT and MRI for Pre-Operative Cochlear Imaging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Abdel-Tawab Mohamed, Principal investigator, Assiut University
Other Study IDs: Imaging in Cochlear implant
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Hearing Loss, Sensorineural
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Tomography, X-Ray Computed; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- "cochlear implantation" group: "cochlear implantation" group: patients undergoing cochlear implantation between December 2019 and December 2021in the ENT department of Assiut university hospital.
  Interventions: Diagnostic Test: Computed Tomography and Magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: Computed Tomography and Magnetic resonance imaging — Preoperative imaging for patients undergoing cochlear implants

SUMMARY:
This study investigates the role of the preoperative computed tomography (CT) and magnetic resonance imaging (MRI) before cochlear implants and their role in selecting suitable patients for surgery.

DETAILED DESCRIPTION:
Cochlear implant is the treatment of choice for deep sensorineural hearing loss, notably in those patients for whom conventional amplification devices do not provide significant clinical improvement. Imaging plays an important role in the workup of cochlear implant candidates not only to identify inner ear congenital and acquired abnormalities or cochlear nerve anomalies but also to detect temporal bone abnormalities that may be encountered during surgery and may alter surgical approach.

Some variations are potential surgical hazards that may lead to problems during the surgery and may alert the surgeon regarding potential surgical dangers and complications.

The radiologist and surgeon must be familiar with these imaging findings. Both computed tomography and magnetic resonance imaging should be used as they delineate, in different manners, cochlear and middle ear anatomy as well as other anatomical variants.

Mastoid pneumatization is important for planning the surgery. It is classified into pneumatic, diploic, sclerotic, and mixed. Effusion of the middle ear cleft should also be reported.

Korner's septum divides the mastoid process into a superficial squamous portion and a deep petrous portion. It may mislead the surgeon to the mastoid antrum during surgery. Mastoid emissary veins participate in extracranial venous drainage of the posterior fossa dural sinuses. Most of them disappear, however, some persist and enlarge.

Low lying dura represents difficulty to access the aditus, lateral semicircular canal, and posterior tympanotomy. It is often associated with sclerotic mastoid. Posterior tympanotomy is a well known otologic procedure that allows surgeons to access the middle ear cavity. The surgeon opens a window in the posterior wall of the middle ear in the angle between the chorda tympani and the mastoid part of the facial nerve. Laterally or anteriorly positioned mastoid part of the facial nerve may hinder the access to the facial recess or may even force the surgeon to change his approach.

The sigmoid sinus passes along the posteromedial border of the mastoid air cells. An anteriorly located sinus produces a deep bulge in the mastoid and may reach the posterior wall of the external auditory canal being separated from it only by a thin bony plate.

Jugular bulb variations are common, the roof of a normal jugular bulb lies either at or slightly below the level of the external auditory canal floor and is separated from the middle ear cavity by the thin bony sigmoid plate. The average width of the jugular bulb is 1 cm. A jugular bulb larger than 1 cm is called a giant or mega jugular bulb. A jugular bulb that extends over the basal turn of the cochlea or abuts the round window is called a high riding jugular bulb. Dehiscence of the sigmoid plate with upward protrusion of the bulb into the posterior hypotympanum is called a dehiscent jugular bulb, which may obliterate a round window niche.

The aberrant internal carotid artery is an enlarged inferior tympanic artery that occurs as a result of agenesis or underdevelopment of the cervical segment of the internal carotid artery. It runs along the medial aspect of the middle ear coursing anteriorly across the cochlear promontory to join the horizontal carotid canal through a dehiscence in the carotid plate.

Cochlear duct patency and axis, patency of the round window niche and the patent even caliber of the cochlea must be adequately evaluated by both computed tomography and magnetic resonance imaging. Otospongiotic foci compromise the insertion of the cochlear implant electrode if they occlude the round window niche or cochlear duct. Labyrinthitis ossificans may partially or completely obliterate cochlear lumen. Fibrosis may precede ossification and areas of fibrosis and ossification may coexist. Cochlear ossification with luminal obstruction is not a contraindication for implantation, however, it is important to be identified preoperatively.

Vestibular aqueduct (VA) is considered dilated if its width is greater than the width of the posterior SCC or if its midpoint width is greater than 1.5 mm. Computed tomography shows dilatation of the VA only whereas magnetic resonance imaging shows the dilatation of the VA and of the endolymphatic sac.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilled criteria for cochlear implant including audiological criteria (as bilateral profound hearing loss not benefiting from hearing aid) and phoniatric criteria as IQ (using Stanford Binet intelligence scale) more than 80 with no medical, surgical, or radiological contraindication for surgery
* Family motivation and commitment for audiologic and phoniatric rehabilitation and follow up
* Confirmation of the presence of cochlear nerve using preimplant MRI.

Exclusion Criteria:

* Patient who did not fulfill the criteria for indicating cochlear implant surgery
* Patients with no records of preoperative investigations
* Patients with major dysplasia or aplasia of the cochlea as a common cavity.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will be performed in Assiut University Hospital, Department of Radiology during the period from May 2019 to May 2021, and will include 50 patients from different age groups and both sex who will be clinically diagnosed as having severe to profound SNHL and fulfill the criteria for the cochlear implant.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Identifying contraindications for cochlear implant | Day 0
  Identifying contraindications for cochlear implant including
  * cochlear nerve aplasia (evidenced by MRI)
  * cochlear and/or labyrinthine aplasia
  * absence of the internal auditory canal and of the petrous apex bone
  * absence or fusion of the ossicles

CONTACTS AND LOCATIONS:
Overall Officials: Abdelkarim H Abdallah, Professor, Study Chair — Assiut University; Hazem A Yousef, MD, Study Director — Assiut University; Reham A Mahmoud, MD, Study Director — Assiut University; Mohamed A Mohamed, MD, Principal Investigator — Assiut University; Mohamed Salah sadek Ibrahim, Master, Study Director — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Digge P, Solanki RN, Shah DC, Vishwakarma R, Kumar S. Imaging Modality of Choice for Pre-Operative Cochlear Imaging: HRCT vs. MRI Temporal Bone. J Clin Diagn Res. 2016 Oct;10(10):TC01-TC04. doi: 10.7860/JCDR/2016/18033.8592. Epub 2016 Oct 1. PMID 27891421
- [Background] Trimble K, Blaser S, James AL, Papsin BC. Computed tomography and/or magnetic resonance imaging before pediatric cochlear implantation? Developing an investigative strategy. Otol Neurotol. 2007 Apr;28(3):317-24. doi: 10.1097/01.mao.0000253285.40995.91. PMID 17414036
- [Background] Westerhof JP, Rademaker J, Weber BP, Becker H. Congenital malformations of the inner ear and the vestibulocochlear nerve in children with sensorineural hearing loss: evaluation with CT and MRI. J Comput Assist Tomogr. 2001 Sep-Oct;25(5):719-26. doi: 10.1097/00004728-200109000-00009. PMID 11584231
- [Background] Jallu AS, Jehangir M, Ul Hamid W, Pampori RA. Imaging Evaluation of Pediatric Sensorineural Hearing Loss in Potential Candidates for Cochlear Implantation. Indian J Otolaryngol Head Neck Surg. 2015 Dec;67(4):341-6. doi: 10.1007/s12070-015-0819-6. Epub 2015 Jan 7. PMID 26693449